CLINICAL TRIAL: NCT00039572
Title: A Phase I/II Trial For Neutron Capture Therapy In Glioblastoma Multiforme And Intracranial Melanoma
Brief Title: Boron Neutron Capture Therapy in Treating Patients With Glioblastoma Multiforme or Melanoma Metastatic to the Brain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BIDMC-E-010284FB; CDR0000069398 (Registry Identifier: PDQ (Physician Data Query)); NEDH-E-010284FB; NCI-V02-1702
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2002-07

CONDITIONS: Brain and Central Nervous System Tumors; Melanoma (Skin); Metastatic Cancer
Keywords: adult glioblastoma; stage IV melanoma; tumors metastatic to brain; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Melanoma; Neoplasm Metastasis; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — 4-boronophenylalanine-fructose

INTERVENTIONS:
Drug: boronophenylalanine-fructose complex

SUMMARY:
RATIONALE: Radiation therapy such as boron neutron capture therapy may kill tumor cells without harming normal tissue.

PURPOSE: Phase I/II trial to study the effectiveness of boron neutron capture therapy in treating patients who have glioblastoma multiforme or melanoma metastatic to the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the time course, uniformity, and severity of acute and chronic normal tissue reactions in patients with glioblastoma multiforme or intracranial melanoma treated with boronophenylalanine-fructose complex (BPA-f) followed by cranial neutron irradiation using a new fission converter beam facility.
* Determine the maximum tolerated dose of cranial neutron capture therapy in these patients.
* Determine, through serial objective measurements, the clinical response in patients treated with this therapy.
* Determine the pharmacokinetics of BPA-f in these patients.

OUTLINE: This is a dose-escalation study of cranial neutron capture therapy (NCT).

Patients receive boronophenylalanine-fructose complex IV over 90 minutes followed by cranial NCT on days 1 and 2.

Cohorts of 3-6 patients receive escalating doses of NCT until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at the MTD.

Patients are followed at 1, 2, 4, 6, 9, and 12 months and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 16 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme OR
* Radiographically diagnosed brain metastases after a diagnosis of melanoma
* Contrast-enhanced tumor volume must not exceed 60 mL

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 6 months

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Creatinine normal

Cardiovascular:

* No prior severe cardiac disease, including the following:

  * Uncontrolled arrhythmias or conduction defects
  * Unstable or newly diagnosed angina pectoris
  * Recent coronary artery disease
  * Congestive heart failure

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after study
* No prior phenylketonuria
* No cognitive impairment that would preclude informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior cranial irradiation

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-05; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M. Busse, MD, PhD, Study Chair — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts Institute of Technology, Cambridge, Massachusetts